CLINICAL TRIAL: NCT05207579
Title: Psychometric Analysis of Urdu Version of Shoulder Pain and Disability Index: A Reliability and Validity Study
Brief Title: Urdu Version of Lower Extremity Functional Scale: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0294
Record Dates: First submitted 2022-01-24; First posted 2022-01-26 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Musculoskeletal Disorder
Keywords: Lower Extremity Functional Scale; Musculoskeletal Disorder; Cultural adaptation; Validity; Urdu Version; Reliability; Lower Extremity
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the research is to translate and to culturally familiarize the Lower extremity functional scale into the Urdu language along the investigation if the Lower Extremity Functional Scale is reliable and validate in the Pakistani population with Lower extremity musculoskeletal disorders and to check the correlation with Short Form - 36.

DETAILED DESCRIPTION:
The questionnaire will be translated into Urdu and cross-culturally modified. Internal consistency, test-retest reliability, conceptual validity, discriminative validity, responsiveness, and concurrent validity will be examined in 150 participants seeking treatment for lower extremity dysfunction using the Urdu version of the Lower Extremity Functional Scale.

ELIGIBILITY:
Inclusion Criteria:

* From16 years Old to 60 Years Old
* Presence of an Lower extremity musculoskeletal disorders like soft tissue injuries, joints and muscles injuries
* No intervention between the test-retest assessments

Exclusion Criteria:

* To complete the forms because of a psychological Impairment.
* Illiteracy or lack of understanding of Urdu Language
* The presence of any kind of bone fracture

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pakistani population with Lower extremity musculoskeletal disorders was included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale | 1st day
  Lower Extremity Functional Scale is a valid and reliable instrument to determine the functional status for acute and chronic lower extremity musculoskeletal dysfunction due to the importance of evidence-based health care
Short Form-36 | 1st day
  Short Form-36 is one of the most widely used and evaluated generic health-related quality of life questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No